CLINICAL TRIAL: NCT00617513
Title: A Double-Blind Placebo-Controlled Dose-Finding Trial to Evaluate the Efficacy and Safety of R093877 in Patients With Chronic Idiopathic Constipation
Brief Title: Efficacy and Safety Study of Prucalopride for the Treatment of Chronic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRU-INT-1
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator)
  Interventions: Drug: Prucalopride
- 2 (Active Comparator)
  Interventions: Drug: Prucalopride
- 3 (Active Comparator)
  Interventions: Drug: Prucalopride
- 4 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Prucalopride — 0.5 mg once daily
  Other Names: Resolor
  Arms: 1
Other: Placebo — o.d.
  Arms: 4
Drug: Prucalopride — 1 mg o.d.
  Other Names: Resolor
  Arms: 2
Drug: Prucalopride — 2 mg o.d.
  Other Names: Resolor
  Arms: 3

SUMMARY:
The purpose of this study is to determine which dose of prucalopride is safe and effective in patients with chronic idiopathic constipation.

Hypothesis:

Prucalopride 1 and 2 mg are safe and effective for the treatment of chronic idiopathic constipation whereas 0,5 mg is a suboptimal dose.

DETAILED DESCRIPTION:
This is a phase II trial with a parallel-group design, consisting of a drug-free run-in phase (phase 1), followed by a placebo controlled double-blind phase (phase 2). Patients will receive either R093877 0.5 mg o.d., 1 mg o.d. or 2 mg o.d. or placebo for a period of 4 weeks.

Phase 1 is a run-in period of 4 weeks duration, during which the bowel habit is documented and the existence of constipation confirmed. At the start of this period all existing laxative medication is withdrawn but patients will be instructed not to change their dietary habits, in particular their fibre intake during the trial. Patients will enter the double-blind phase if constipation has been shown to be present during the run-in period.

If the definition of constipation was not met during the 4 weeks of the run-in period, double-blind treatment will not be started.

Phase 2 is a double-blind, randomized, placebo-controlled phase, in which patients will be treated for 4 weeks with either 0.5 mg, 1 mg or 2 mg of R093877 or placebo given once daily (one capsule is taken before breakfast).

Patients admitted to the double blind treatment period will be randomly allocated to one of the 4 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years.
* History of constipation i.e., the patient reported the occurrence of TWO OR MORE of the following criteria for at least 6 months before the selection visit :

  1. two or fewer spontaneous* bowel movements in a week.
  2. lumpy (scyballae) and/or hard stools at least a quarter of the stools.
  3. sensation of incomplete evacuation following at least a quarter of the stools.
  4. straining at defaecation at least a quarter of the time. *A bowel movement was considered spontaneous if it was not preceded by the intake of a laxative agent within a period of 12 hours. An amendment was made changing this period to 24 hours. Moreover, the amendment stated: "Patients who never opened their bowels spontaneously would be considered constipated and eligible to enter the double-blind phase of the trial, whether or not the above mentioned criteria were met for laxativa/enemas induced stools".
* Constipation causing disability; the patient's occupational, social and recreational activities were governed by his/her constipation and efforts to attain relief.
* Normal electromyographic inhibition pattern of the external anal sphincter during straining (clinical and/or electromyographic and/or manometric evidence is acceptable).
* Absence of organic abnormalities of the colon on barium enema or on total colonoscopic examination. This criterion was amended to: "If complaints of constipation were of recent onset,i.e., had been present for 6 months to 1 year, results of a colonoscopic examination performed within the last 12 months were needed. If complaints of constipation had been present for more than one year, results of an endoscopic examination performed within the past three years were acceptable".
* Poor results with laxative treatment and diet counselling.
* Constipation of a functional, i.e., idiopathic nature.
* Availability of the patient's written informed consent.
* Patient available for follow-up during the trial period as determined in the protocol.

Exclusion Criteria:

* Constipation thought to be drug-induced.
* Presence of secondary causes of constipation, for instance: endocrine disorders, metabolic disorders, neurologic disorders.
* Congenital megacolon/megarectum.
* History of previous abdominal surgery other than hysterectomy, surgery for Meckel's diverticle,appendicectomy, cholecystectomy, inguinal repair, splenectomy, nephrectomy or fundoplication.
* Known or suspected organic disorders of the large bowel, i.e., obstruction, carcinoma or inflammatory bowel disease.
* Active proctological conditions which were thought to be responsible for constipation.
* Evidence of a non-relaxing pelvic floor ("anismus") as the main cause of constipation.
* Clinically significant ECG abnormalities.
* Known illnesses or conditions which might interfere in any way with the adequate assessment of the drug under study, such as severe cardiovascular or lung disease, neurologic or psychiatric disorders, alcoholism, cancer or AIDS.
* Impaired renal function
* Presence of a serum amylase-, a serum glutamic-oxaloacetic transaminase (SGOT) or a serum glutamic-pyruvic transaminase (SGPT) concentration of > 2 times the upper limit of normal.
* Clinically significant abnormalities of blood chemistry, haematology or urinalysis at selection.
* Pregnancy or wish to become pregnant during the course of the study. - Breast feeding.
* Investigational drug received in the 30 days preceding the trial.
* Known use of street drugs e.g., marijuana, cocaine etc.
* Unability or unwillingness to return for required follow-up visits.
* Reliability and physical state preventing proper evaluation of a drug trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 1995-03; Primary Completion 1996-03 (Actual); Study Completion 1996-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of prucalopride and to compare the effects of 0.5 mg, 1 mg or 2 mg of R093877 versus placebo | 4 weeks

SECONDARY OUTCOMES:
Evaluation of the effects of R093877 on symptoms associated with idiopathic constipation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc Van Outryve, MD, Principal Investigator — Jan Palfijn Hospital

REFERENCES:
- [Derived] Emmanuel A, Cools M, Vandeplassche L, Kerstens R. Prucalopride improves bowel function and colonic transit time in patients with chronic constipation: an integrated analysis. Am J Gastroenterol. 2014 Jun;109(6):887-94. doi: 10.1038/ajg.2014.74. Epub 2014 Apr 15. PMID 24732867